CLINICAL TRIAL: NCT04486417
Title: Feasibility of a Telematics Pre-operative Assessment in a Bariatric Center of Excellence During Covid-19 Phase 2: a Prospective Observational Study
Brief Title: Feasibility of a Telematics Pre-operative Assessment in a Bariatric Surgery During Covid-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianfranco Silecchia, Full Professor, University of Roma La Sapienza
Other Study IDs: 66.20
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-06

CONDITIONS: Obesity; Telemedicine; Bariatric Surgery
Keywords: Bariatric Surgery; Telemedicine; Covid-19; Pre-operative psychological assessment; Pre-operative nutritional counseling
MeSH Terms: conditions — Obesity; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronavirus (COVID-19) is a respiratory disease caused by a newly discovered coronavirus, SARS-CoV-2. Several recent papers on the pandemic recognized obesity as a risk factor for the COVID-19 infection. Therefore, an effective treatment for obesity even during COVID-19 outbreak is needed. Bariatric surgery, is considered an effective treatment in the reduction of obesity-related comorbidities and mortality risk. However, during Covid-19 phase 1 (lockdown) the near totality of elective non-oncologic procedures, including bariatric surgery, has been postponed, and all the outpatients' visits too. Therefore, phase 1 led to completely change the way of managing the pre-operative multidisciplinary visits considering the hospital limitation access and the restriction. In the present study the investigators explored the use of telemedicine as a possible strategy to face this new situation.

Specifically, this study aims to test the efficacy of an online structured protocol based on pre-operative multidisciplinary assessment using telemedicine instruments. In particular, the primary end point is to test the feasibility of a telematics pre-operative work-up. The secondary end points are evaluating patient's compliance and satisfaction to the online assessment.

DETAILED DESCRIPTION:
Coronavirus (COVID-19) is a respiratory disease caused by a newly discovered coronavirus, SARS-CoV-2. In Italy the first person-to-person transmission was reported on February, 21, 2020. The North of Italy, became the epicentre of the outbreak in Europe, and Italy was one of the most affected Country in the World. As May, 5, 2020 the total number of positive Covid-19 in Italy was 212532, with 27400 deaths. Several recent papers on the pandemic recognized obesity as a risk factor for the COVID-19 infection. Furthermore, the Centre for Disease and Control Prevention report that people with diabetes, liver disease, chronic lung disease and cardiovascular disease are at higher risk for greater severity of COVID-19, and these are the most common obesity-related comorbidities too. In New York out of 3615 subjects with SARS-CoV-2 positive swab between March 4, and April 4, 21% had BMI 30-34 and 16% had BMI > 35.

This foreword underlines the need to guarantee gold standard treatment for obesity even during COVID-19 outbreak, including bariatric surgery, considered an effective treatment in the reduction of obesity-related comorbidities and mortality risk.

On March 9, 2020 started the phase 1 (lockdown) and the near totality of elective non-oncologic procedures has been postponed (including bariatric procedures) to increase capacity for in-patient beds and acute care.

The efforts during the unexpected and unexplored phase 1 were addressed how to properly prepare the phase 2, started on May,4, 2020. In fact, the Phase 1 led to completely change the way of managing the pre-operative multidisciplinary outpatient's visits considering the hospital limitation access and the restriction.

All the possible remote contact with patients has been explored, in order to face this new situation. The first challenge was: how to continue to support our patients seeking treatment of morbid obesity. Considering the lack of effective treatment for Covid-19 and the possibility of a new epidemic peak, new strategies to assess and treat morbid obesity patients are needed.

Among possible strategies telemedicine could be the answer. Previous studies showed the efficacy of telemedicine (telephone or videoconferences) in bariatric surgery treatment, but no studies have ever tested a structured protocol during the Covid-19 pandemic, even if it is strongly encouraged according to recent suggestions of scientific community in bariatric field.

This study aims to test the efficacy of an online structured protocol based on pre-operative multidisciplinary assessment using telemedicine instruments.

In particular, the primary end point is to test the feasibility of a telematics pre-operative work-up. The secondary end points are evaluating patient's compliance and satisfaction to the online assessment.

Materials and Methods Participants The protocol will be tested on 20 patients of the Bariatric Center of Excellence, "Sapienza" University of Rome. All patients, whose first contact was at the hospital before the lockdown for the surgical session, will be contacted starting from the booking list. Each patient will be contacted by phone in order to be informed about the online assessment procedure and to ask for consent.

Protocol The protocol consists in a three weekly one-to-one online sessions both for nutritional and psychological pre-operative assessment, using skype or whatsapp, and a face to face session (psychological, nutritional and surgical) for the final decision on the bariatric surgery suitability. The standard related to privacy, informed consent and setting will respect the more recent guidelines for online consultations.

The nutritional sessions will be structured as follow:

1. a) Session 1 (30 minutes) All the patients will be previously instructed by telephone to collect a centimetre and a weighing scale to take the anthropometric measures and weight.

   During the first session the following data will be collected: weight history, previous diets attempts, physical activity and lifestyle habits, food intake modality (greed, chewing and distribution of meals), water intake, evacuation. In order to detect food intake and eating habits, a 7-days food diary will be explained and sent to the patients by email with an instruction sheet. One week later the patient will send the diary back.

   In session 1 anthropometric measures (body weight, waist and hip circumferences and referred height) will be collected: height and weight will be used to calculate body mass index (BMI) in order to categorize patient's obesity level. The patient will send a picture of the weight by e-mail, instead circumferences will be taken following the dietician's instruction, who observe through the video.
2. a) Session 2 (30 minutes) A week later the patient will send the 7-days food diary and picture of the daily weight by e-mail. The dietician will work on the food diary focusing on the wrong eating habits and choices. Then a customized food plan will be created (Low Calorie Diet or Very Low Calorie Diet or Very Low Calorie Ketogenic Diet) in order to be followed for the next 2 weeks. The Very Low Calorie Ketogenic Diet will be prescribed in high risk patients. Than, will be asked to complete a new 7-days food diary and to send it back in 2 weeks. In addition, a physical activity program will be prescribed.
3. a) Session 3 (30 minutes) After 14 days of diet, the patient's weight and the 7-days food diary will be collected and discussed. The dietician and the patient will also discuss on the reached results comparing with those expected in 3 sessions. Level of compliance to recommendations will be evaluated in order to proceed at the final session.

The psychological sessions will be structured as follow:

1. b) Session 1 (50 minutes' interview + 40 minutes' psychometric questionnaires administration) During the first session psychological anamnesis (previous and recent psychopathological symptoms, somatic signs, any psychiatric or neurological pharmacotherapies, history of psychotherapies, significant life events, familiar psychopathology), life history, family structure and relations will be collected following National guidelines. The replicable online version of some psychometric questionnaires will be administered; in particular, Binge Eating Scale (BES) and Eating Attitude Test - 26 (EAT-26) to assess eating disorders, Hamilton for Depression (HAM-D) and Anxiety (HAM-A) to assess mood disorders, SIO- Obesity correlated Disability Test to assess quality of life. All questionnaires will be created using "google moduli", and the generated link to access to the online questionnaire will be sent to the patients by e-mail. The answers will be automatically uploaded on an excel sheet combined with "google moduli" questionnaire sheet. The administration will follow APA guidelines on psychological tele-assessment.
2. b) Session 2 (50 minutes) In the second session the psychologist will discuss the questionnaires' results. Than, information on weight history and possible related significant life events, expectations on weight loss after surgery, motivation, and compliance to previous treatment will be collected.
3. b) Session 3 (50 minutes) All the detected data, including compliance to nutritional recommendation and reached weight loss will be considered. The psychologist summarized the sessions 'contents, and discussed on the future expectation and changes after surgery. Level of compliance will be evaluated in order to proceed to the final session.

4) Final multidisciplinary session - one-to-one modality Respecting the interpersonal safety distance and all the recommended indications of phase 2 measures, final multidisciplinary sessions (psychological, nutritional and surgical) will be carried out at the hospital. All the team members will previously discuss each case, each possible online session observed problems, patients 'compliance and reached results compared to expected. Than, psychologist and dietician will carry on the one-to-one last session, discussing on patient's suitability/non suitability to surgery (according to the procedural guideline), and on all the steps to comply with (eg. diet changes, follow up timing, expected possible inconveniences or difficulties).

Expected results Less than 20% of rejection rate to the online assessment request and an high rate of continuation until the end of the assessment are expected. Furthermore, more than 50% of patients are expected to be compliant and satisfied with the online procedure.

ELIGIBILITY:
Inclusion Criteria:

* not being positive to Covid-19 (according to Covid-19 telephone interview)
* age >18 and <65 years
* availability of a stable internet connection
* having a mailbox and possibility to send and receive pdf documents via e-mail

Exclusion Criteria:

* Not having a stable internet connection and a mailbox
* not having practicality with telematic tools
* having possible Covid-19 symptoms (according to Covid-19 telephone interview)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese people asking for bariatric surgery, who are in the waiting list of the bariatric center
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-07-22 (Actual); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Rejection rate (%) | During the recruitment process
  The rejection rate to the online assessment modality will be calculated (% of people who refuse to participate to the online assessment procedure).
Drop out rate | 1 month
  The drop out rate will be calculated (% of people who drop out during the assessment procedure)

SECONDARY OUTCOMES:
Excess Weight Loss percentage (EWL%) | 1 month
  The patient's compliance to the clinicians' indications will be evaluated considering an Excess Weight Loss (%) >=5% for each participant, which will be calculated according to this formula: 100% × (weight at session 1 - weight at session 4)/(weight at session 1 - ideal body weight). The percentage of people with an EWL>=%5 will be reported.
Satisfaction degree | 3 weeks
  A questionnaire on satisfaction degree was specifically created. It asked to participants the following questions:
  * Are you satisfied with the psychological and nutritional online assessment? YES/NO
  * Which was your level of satisfaction with the online assessment? from 0 to 10 (where 0 = not at all, 10 = very much)
  * How would you rate the quality of video calls? from 0 to 10 (where 0 = not of quality (I couldn't see/hear at all; ) 10 = excellent quality (I could see/hear well))
  * In your opinion, could an online pre-operative psychological and nutritional assessment be effective? YES/NO
  * Would you have preferred to carry out the psychological and nutritional assessment in person? YES/NO
  * Was it difficult to use electronic tools for filling in / sending questionnaires? YES/NO
  * In light of this pre-operative online evaluation, would you carry out post-operative psychological and nutritional follow-up using videocalls? YES/NO

CONTACTS AND LOCATIONS:
Locations (1):
- Gianfranco Silecchia, Latina, Italy

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Zheng KI, Gao F, Wang XB, Sun QF, Pan KH, Wang TY, Ma HL, Chen YP, Liu WY, George J, Zheng MH. Letter to the Editor: Obesity as a risk factor for greater severity of COVID-19 in patients with metabolic associated fatty liver disease. Metabolism. 2020 Jul;108:154244. doi: 10.1016/j.metabol.2020.154244. Epub 2020 Apr 19. No abstract available. PMID 32320741
- [Background] Caussy C, Wallet F, Laville M, Disse E. Obesity is Associated with Severe Forms of COVID-19. Obesity (Silver Spring). 2020 Jul;28(7):1175. doi: 10.1002/oby.22842. Epub 2020 May 21. No abstract available. PMID 32314861
- [Background] Lighter J, Phillips M, Hochman S, Sterling S, Johnson D, Francois F, Stachel A. Obesity in Patients Younger Than 60 Years Is a Risk Factor for COVID-19 Hospital Admission. Clin Infect Dis. 2020 Jul 28;71(15):896-897. doi: 10.1093/cid/ciaa415. No abstract available. PMID 32271368
- [Background] Andolfi C, Fisichella PM. Epidemiology of Obesity and Associated Comorbidities. J Laparoendosc Adv Surg Tech A. 2018 Aug;28(8):919-924. doi: 10.1089/lap.2018.0380. Epub 2018 Jul 16. PMID 30010474
- [Background] Nguyen NT, Varela JE. Bariatric surgery for obesity and metabolic disorders: state of the art. Nat Rev Gastroenterol Hepatol. 2017 Mar;14(3):160-169. doi: 10.1038/nrgastro.2016.170. Epub 2016 Nov 30. PMID 27899816
- [Background] Coldebella B, Armfield NR, Bambling M, Hansen J, Edirippulige S. The use of telemedicine for delivering healthcare to bariatric surgery patients: A literature review. J Telemed Telecare. 2018 Dec;24(10):651-660. doi: 10.1177/1357633X18795356. PMID 30343656
- [Background] Zhang MW, Ho RC, Cassin SE, Hawa R, Sockalingam S. Online and smartphone based cognitive behavioral therapy for bariatric surgery patients: Initial pilot study. Technol Health Care. 2015;23(6):737-44. doi: 10.3233/THC-151026. PMID 26409514
- [Background] Yeo C, Ahmed S, Oo AM, Koura A, Sanghvi K, Yeo D. COVID-19 and Obesity-the Management of Pre- and Post-bariatric Patients Amidst the COVID-19 Pandemic. Obes Surg. 2020 Sep;30(9):3607-3609. doi: 10.1007/s11695-020-04670-6. No abstract available. PMID 32385668
- [Background] McEneaney DF, Lennie SC. Video instructions improve accuracy of self-measures of waist circumference compared with written instructions. Public Health Nutr. 2011 Jul;14(7):1192-9. doi: 10.1017/S1368980011000450. Epub 2011 Mar 31. PMID 21450137
- [Background] Fried M, Hainer V, Basdevant A, Buchwald H, Deitel M, Finer N, Greve JW, Horber F, Mathus-Vliegen E, Scopinaro N, Steffen R, Tsigos C, Weiner R, Widhalm K. Interdisciplinary European guidelines on surgery of severe obesity. Obes Facts. 2008;1(1):52-9. doi: 10.1159/000113937. Epub 2008 Feb 8. PMID 20054163
- [Background] Garner DM, Olmsted MP, Bohr Y, Garfinkel PE. The eating attitudes test: psychometric features and clinical correlates. Psychol Med. 1982 Nov;12(4):871-8. doi: 10.1017/s0033291700049163. PMID 6961471
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Hamilton M. Development of a rating scale for primary depressive illness. Br J Soc Clin Psychol. 1967 Dec;6(4):278-96. doi: 10.1111/j.2044-8260.1967.tb00530.x. No abstract available. PMID 6080235
- [Background] Donini LM, Brunani A, Sirtori A, Savina C, Tempera S, Cuzzolaro M, Spera G, Cimolin V, Precilios H, Raggi A, Capodaglio P; SIO-ISDCA Task Force. Assessing disability in morbidly obese individuals: the Italian Society of Obesity test for obesity-related disabilities. Disabil Rehabil. 2011;33(25-26):2509-18. doi: 10.3109/09638288.2011.575529. Epub 2011 May 4. PMID 21542694
- See also: American Psychological Association (2020). Guidance on psychological tele-assessment during the COVID-19 crisis. Accessed 7 May 2020 — https://www.apaservices.org/practice/reimbursement/health-codes/testing/tele-assessment-covid-19
- See also: Società Italiana di Chirurgia dell'obesità (SICOb). Linee guida di chirurgia dell'obesità. Accessed 7 May 2020 — https://www.sicob.org/00_materiali/linee_guida_2016.pdf
- See also: Società Italiana di Nutrizione Umana (SINU). (2014). Livelli di Assunzione di Riferimento di Nutrienti ed energia per la popolazione italiana IV Revisione (LARN 2014). Accessed 7 May 2020 — https://sinu.it/tabelle-larn-2014/